CLINICAL TRIAL: NCT05683912
Title: Aflibercept for Diabetic Macular Edema In Real-life Practice in GREece: The ADMIRE Study
Brief Title: Aflibercept for Diabetic Macular Edema In Real-life Practice in GREece
Acronym: ADMIRE
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Irini Chatziralli, Assistant Professor in Ophthalmology, University of Athens
Other Study IDs: 698/2019
Record Dates: First submitted 2022-12-27; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Aflibercept — Intravitreal aflibercept as used in the routice clinical practice

SUMMARY:
ADMIRE was a prospective, observational cohort study of patients with diabetic macular edema (DME). Efficacy was assessed by change in best-corrected visual acuity (BCVA) and central retinal thickness (CRT) from baseline to months 12, 24 and 36 after treatment with intravitreal aflibercept in treatment-naïve patients and previously treated patients. Safety was evaluated by recording any patients-reported events.

ELIGIBILITY:
Inclusion Criteria:

Patients with DM, able to give written informed consent Patients with DME>320 μm, who need treatment

Exclusion Criteria:

Patients with other retinal diseases than DME Intraocular surgery within the last 6 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DME treated with intravitreal aflibercept 2.0mg in routice clinical practice.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No